CLINICAL TRIAL: NCT03206944
Title: Antiplatlet Effects of Standardized Tomato Extract in Hypertensive Subjects at High Estimated Cardiovascular Risk
Brief Title: Antiplatlet Effects of Standardized Tomato Extract in Hypertensive Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beata Krasinska (Other)
Responsible Party: Sponsor-Investigator, Beata Krasinska, Principal Investigator, Poznan University of Medical Sciences
Organization: Poznan University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 377/2015
Record Dates: First submitted 2017-06-27; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Hypertension,Essential; Obesity
Keywords: standardized tomato extract; anti-aggregation; high cardiovascular risk; diet supplement
MeSH Terms: conditions — Essential Hypertension; Obesity | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 ASA (Experimental): Group 1(ASA) included 33 patients who received acetylsalicylic acid at a dose of 75 mg orally once a day in the morning.
  Interventions: Drug: acetylsalicylic acid
- Group 2 STE (Experimental): Group 2 (STE) included 32 patients receiving tomato fruit extract (STE) (ZAAX, Sequia, Poland) at a dose of 213 mg orally once a day in the morning.
  Interventions: Drug: Tomato Fruit Extract

INTERVENTIONS:
Drug: acetylsalicylic acid — Group 1(ASA) included 33 patients who received acetylsalicylic acid at a dose of 75 mg in the morning
  Other Names: Group 1 ASA
  Arms: Group 1 ASA
Drug: Tomato Fruit Extract — Group 2 (STE) included 32 patients receiving standardized tomato extract (STE) (ZAAX, Sequia, Poland) at a dose of 213 mg orally in the morning
  Other Names: Group 2 STE
  Arms: Group 2 STE

SUMMARY:
The reducing the anti-aggregation properties of platelets significantly decreases the risk of myocardial infarction and the total number of cardiovascular events. In patients who have cardiovascular disease, anti-platelet therapy reduces the risk of serious vascular events. Side effects, such as bleeding, are relatively small so the benefits of anti-platelet therapy in secondary prevention exceed the risk of these side effects. According to guidelines for the treatment of arterial hypertension, PTNT 2015, patients with arterial hypertension (HA) that have a 20% or higher risk for cardiovascular events in the next 10 years, should have ASA included in their treatment to reduce this risk. It has been proved that the use of acetylsalicylic acid in secondary prevention reduces the risk of major cardiovascular events, while the benefits of ASA in primary prevention have recently been debated. The benefits of using ASA in primary prevention should always be confronted with the risk of hemorrhagic complications of this therapy According to 2016 European Guidelines on cardiovascular disease (CVD) prevention in clinical practice, anti-platelet therapy is not recommended in individuals who do not suffer from CVD, due to the increased risk of major bleeding. It is important to look for alternative anti-platelet therapy for people with cardiovascular risk factors. Standardized tomato extract (STE) does not cause side effects and may have multiple beneficial effects on total cardiovascular risk, primarily by inhibiting platelet aggregation. Since its discovery in 1999, several studies and human trials with STE have been carried out. During the last 50 years, tomato (Lycopersicon esculentum) has become a highly consumed food. The benefits of inhibiting platelet activity through diet are currently difficult to determine due to the lack of clear and comprehensive scientific data. It is difficult to specify the over activity of the plaques or their proper activity. However, there are data available that indicate the benefits of a diet containing diminishing activity of platelets (Mediterranean diet) and lowering cardiovascular risk.The investigators want to conduct a comparison of the less common STE with clinically recognized ASA. The aim of the study was to compare the anti-platelet effect of STE and ASA in hypertensive patients with high cardiovascular risk.The study highlights that STE may be an alternative, food-based strategy to control the platelets reactivity.

DETAILED DESCRIPTION:
Study design The study involved 82 high-risk hypertensive patients (44 men and 38 women), aged 28-74years, conducted between July 2015 and February 2017 in the Department of Hypertension at the University of Medical Sciences in Poznan. Seventeen patients reported resignation during the study. The permission no. 377/15 to conduct the study was published by the Ethics Committee at the Poznan University of Medical Sciences. All the patients gave informed consent for participation in the study. Patients with primary hypertension and high cardiovascular risk were randomly assigned to one of two groups. Group 1(ASA) included 33 patients who received acetylsalicylic acid at a dose of 75 mg in the morning. Group 2 (STE) included 32 patients receiving standardized tomato extract (STE) (ZAAX, Sequia, Poland) at a dose of 213 mg orally in the morning.

The patients had two visits within 4 weeks according to the scheme:

Visit 1: During the first visit, patients were qualified for the study. The patients with previously diagnosed hypertension were referred from an outpatient clinic, to the hospital ward. After admission, the patients with high cardiovascular risk were isolated and written consents were obtained.

On the basis of stage of hypertension, presence of risk factors and subclinical organ damage, diabetes coexistence, cardiovascular complications and chronic kidney disease the cardiovascular risk was estimated. Each patient with one or two risk factors and a blood pressure (BP) > 180/110 mmHg or three or more risk factors, and a BP >160/100 mmHg or with the presence of organ damage and BP >140/90 mmHg were classified as a high risk Group.There have been no changes in the concomitant treatment (lipid-lowering, anti-hypertensive and antidiabetic) during the study.

Numerous laboratory tests and imaging, such as aldosterone and ARO levels, both before and after tilting, creatinine, urea, GFR, sodium, potassium, pro BNP, TSH, FT3, FT4, and a 24-hour collection for electrolytes were collected. Abdominal ultrasound examinations, computed tomography of the abdomen, and Doppler ultrasound of the renal arteries were performed to exclude secondary causes of hypertension. Clinical BP measurements were performed three times, as well as, ambulatory blood pressure monitoring (ABPM) and echocardiography was conducted. Whole blood samples were taken and baseline platelet aggregation was determined using the VerifyNow analyzer from Accumetrics. In Group 1, two whole blood samples for VerifyNow Aspirin test were assayed. In Group 2, four whole blood samples for VerifyNow Aspirin and P2Y12 tests were assayed.

Visit 2: After 4 weeks of taking STE or ASA the patients visited the hospital for the second visit. All examinations from visit 1, including platelet aggregation inhibition assays, were repeated. Whole blood samples were collected 1-4 h after the ingestion of a morning ASA or STE dose from a peripheral vein using a 21 gauge or larger needle in a partial fill 3.2% citrate vacuum collection tube.

Standarized tomato extract characteristics STE is a water-soluble tomato concentrate, free of lycopene and fats, which contains 37 biologically active compounds of well-known structure. These bioactive compounds contain nucleosides (adenosine, cytidine, guanosine, inosine, AMP, GMP), polyphenols including flavonoids (rutin, quercetin, kemferol, luteoline, naryngenin) and phenolic acids (chlorogenic, coffee, p-coumar, ferulic).

In 2009, the European Food Safety Authority (EFSA) approved the water soluble tomato concentrate (WSTC) as a food supplement which helps to maintain normal platelet aggregation. EFSA recommended the use of STE in healthy individuals between 35 and 70. The effective daily dose was 3 g of bioactive compounds contained in syrup or 65-150 mg in powdered form.

This extract affects the inhibition of ADP-mediated aggregation, thromboxane, collagen, von Willebrand factor, thrombin and inflammatory mediators. What is more, it blocks the P2Y12 receptor for ADP and limits intracellular granular release of thromboxane, ADP, selectin P and factor 4 (PF4, platelet factor 4). Additionally, it prevents activation of αIIbβIII integrin and inhibits (GP) IIb / IIIa receptor activation. By inhibiting the P2Y12 receptor for ADP, it increases cAMP activity and this results in decreasing intracellular calcium ions concentration. Inhibition of collagen binding process with GP VI as well as von Willebrand factor with GP Ib receptor and decrease in Cβ and Cy2 phospholipase activity are also included in anti-aggregation effects of STE. These phenomena affect the shape of thrombocytha and are reversible while maintaining a level of platelet activity that allows aggregation in case of vascular injury. ZAAX can be used by people with hypersensitivity to salicylates and other non-steroidal anti-inflammatory drugs, with bronchial asthma, with active peptic ulceration.

Studies have shown that STE inhibits the activation of endothelial inflammatory processes, which prevents the development of atherosclerosis. STE reduces the production of inflammatory cytokines (TNF-α, IL-1β and IL-12) and to increases the synthesis of interleukin 10, which has anti-inflammatory properties.

VerifyNow® Tests Procedure The study protocol included measurements of platelet reactivity using a VerifyNow Tests Procedure (Accumetrics Inc., USA). This method detects platelet activity by measurement of platelet aggregation, in a blood sample, exposed to a specific agonist. This leads to an inhibition of platelet function in response to anti-platelet therapy. The VerifyNow System is a whole blood device that performs qualitative measurement of induced platelet aggregation based on the increase in light transmittance. Two types of VerifyNow test kits were used in the study: VerifyNow Aspirin Test and VerifyNow P2Y12. The Aspirin test results are reported as Aspirin Reaction Units (ARU), which are calculated as a function of the rate of aggregation. ARU values less than 550 indicate effective result of ASA, while values > 550 ARU indicate no effect of the drug. The VerifyNow P2Y12 test measures platelet function based on the ability of activated platelets to bind fibrinogen and provides information on the aggravation of platelet aggregation in reactivity units of P2Y12 receptor (PRU). It is considered that the range of 95 - 208 PRU is responsible for optimal antiplatelet activity. High PRU values after drug administration, point to the lack of expected anti-platelet effect.

Blood pressure measurements In all the patients, during each visit, BP measurements were performed three times at rest, in the supine position, in standard conditions, and using an upper arm blood pressure monitor (Omron 705IT). Ambulatory, 24-hour blood pressure measurements (ABPM) were carried out using an A&D, 24-hour ambulatory peripheral blood pressure monitor. The frequency of measurements was every 15 minutes between 7:00 and 22:00 and every 30 minutes between 22:00 and 7:00.

Statistical analysis Statistical analyses were performed with Statistica, version 12.5. (StatSoft, USA). Since the tested data did not meet the assumption of Gaussian distribution (evaluated with Shapiro-Wilk method), the non-parametric methods were applied. The Wilcoxon signed-rank test was used for evaluation of the differences between the initial values and the values obtained after the treatment, for factors of; body weight composition, blood pressure, and platelet aggregation. To evaluate differences and correlations between the two independent groups the Mann-Whitney U test and Spearman׳s rank correlation coefficient (Rs) were used, respectively. The data presented on graphs and tables included median and interquartile ranges. A p<0.05 was considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* Primary hypertension

Exclusion Criteria:

* secondary hypertension,
* white coat hypertension,
* coronary artery disease,
* myocardial infarction,
* revascularization,
* stroke,
* TIA,
* lower limb atherosclerosis,
* congestive heart failure NYHA III-IV,
* chronic kidney disease (GFR 30 ml/min),
* addiction to alcohol and psychotropic substances,
* active cancer,
* congenital or acquired haemostatic disorder,
* use of ASA, STE, or other antiplatelet agents within the last 14 days.
* additional ex-clusion criteria for Group 2 were hypersensitivity to acetylsalicylic acid and ac-tive gastric or duodenal ulcers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Inhibition of platelet function in response to anti-platelet therapy STE and ASA | 1 month
  The platelet inhibition after STE and ASA therapy (VerifyNow Aspirin for ASA and STE Groups and VerifyNow P2Y12 for STE Group only) The platelet reactivity measurements will be performed using the VerifyNow Tests (Accumetrics Inc., USA) method.

SECONDARY OUTCOMES:
The reduction in BP after STE therapy | 1 month
  The reduction in office BP (measured three times in standard conditions) and in 24-hour ABPM parameters

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Tykarski, Prof, Study Director — Department oh Hypertension, Angiology and Internal Disease. University of Medical Sciences. Poznan,Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Result] Antithrombotic Trialists' (ATT) Collaboration; Baigent C, Blackwell L, Collins R, Emberson J, Godwin J, Peto R, Buring J, Hennekens C, Kearney P, Meade T, Patrono C, Roncaglioni MC, Zanchetti A. Aspirin in the primary and secondary prevention of vascular disease: collaborative meta-analysis of individual participant data from randomised trials. Lancet. 2009 May 30;373(9678):1849-60. doi: 10.1016/S0140-6736(09)60503-1. PMID 19482214
- [Result] O'Kennedy N, Raederstorff D, Duttaroy AK. Fruitflow(R): the first European Food Safety Authority-approved natural cardio-protective functional ingredient. Eur J Nutr. 2017 Mar;56(2):461-482. doi: 10.1007/s00394-016-1265-2. Epub 2016 Jul 7. PMID 27388464
- [Result] F Piepoli M. 2016 European Guidelines on cardiovascular disease prevention in clinical practice : The Sixth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of 10 societies and by invited experts). Int J Behav Med. 2017 Jun;24(3):321-419. doi: 10.1007/s12529-016-9583-6. No abstract available. PMID 28290077
- [Result] Hu FB, Rimm EB, Stampfer MJ, Ascherio A, Spiegelman D, Willett WC. Prospective study of major dietary patterns and risk of coronary heart disease in men. Am J Clin Nutr. 2000 Oct;72(4):912-21. doi: 10.1093/ajcn/72.4.912. PMID 11010931
- [Result] O'Kennedy N, Crosbie L, van Lieshout M, Broom JI, Webb DJ, Duttaroy AK. Effects of antiplatelet components of tomato extract on platelet function in vitro and ex vivo: a time-course cannulation study in healthy humans. Am J Clin Nutr. 2006 Sep;84(3):570-9. doi: 10.1093/ajcn/84.3.570. PMID 16960171
- [Result] Fuentes E, Forero-Doria O, Carrasco G, Marican A, Santos LS, Alarcon M, Palomo I. Effect of tomato industrial processing on phenolic profile and antiplatelet activity. Molecules. 2013 Sep 17;18(9):11526-36. doi: 10.3390/molecules180911526. PMID 24048285
- [Result] Navarrete S, Alarcon M, Palomo I. Aqueous Extract of Tomato (Solanum lycopersicum L.) and Ferulic Acid Reduce the Expression of TNF-alpha and IL-1beta in LPS-Activated Macrophages. Molecules. 2015 Aug 21;20(8):15319-29. doi: 10.3390/molecules200815319. PMID 26307961
- [Result] Schwager J, Richard N, Mussler B, Raederstorff D. Tomato Aqueous Extract Modulates the Inflammatory Profile of Immune Cells and Endothelial Cells. Molecules. 2016 Jan 29;21(2):168. doi: 10.3390/molecules21020168. PMID 26840280
- [Result] Tektonidis TG, Akesson A, Gigante B, Wolk A, Larsson SC. Adherence to a Mediterranean diet is associated with reduced risk of heart failure in men. Eur J Heart Fail. 2016 Mar;18(3):253-9. doi: 10.1002/ejhf.481. Epub 2016 Jan 18. PMID 26781788
- [Result] Tektonidis TG, Akesson A, Gigante B, Wolk A, Larsson SC. A Mediterranean diet and risk of myocardial infarction, heart failure and stroke: A population-based cohort study. Atherosclerosis. 2015 Nov;243(1):93-8. doi: 10.1016/j.atherosclerosis.2015.08.039. Epub 2015 Sep 3. PMID 26363438
- [Result] Burton-Freeman B, Sesso HD. Whole food versus supplement: comparing the clinical evidence of tomato intake and lycopene supplementation on cardiovascular risk factors. Adv Nutr. 2014 Sep;5(5):457-85. doi: 10.3945/an.114.005231. PMID 25469376
- [Result] Jacques PF, Lyass A, Massaro JM, Vasan RS, D'Agostino RB Sr. Relationship of lycopene intake and consumption of tomato products to incident CVD. Br J Nutr. 2013 Aug 28;110(3):545-51. doi: 10.1017/S0007114512005417. Epub 2013 Jan 15. PMID 23317928
- [Result] Ghavipour M, Saedisomeolia A, Djalali M, Sotoudeh G, Eshraghyan MR, Moghadam AM, Wood LG. Tomato juice consumption reduces systemic inflammation in overweight and obese females. Br J Nutr. 2013 Jun;109(11):2031-5. doi: 10.1017/S0007114512004278. Epub 2012 Oct 15. PMID 23069270
- [Result] Canene-Adams K, Campbell JK, Zaripheh S, Jeffery EH, Erdman JW Jr. The tomato as a functional food. J Nutr. 2005 May;135(5):1226-30. doi: 10.1093/jn/135.5.1226. PMID 15867308
- [Result] Dutta-Roy AK, Crosbie L, Gordon MJ. Effects of tomato extract on human platelet aggregation in vitro. Platelets. 2001 Jun;12(4):218-27. doi: 10.1080/09537100120058757. PMID 11454256
- [Result] O'Kennedy N, Crosbie L, Whelan S, Luther V, Horgan G, Broom JI, Webb DJ, Duttaroy AK. Effects of tomato extract on platelet function: a double-blinded crossover study in healthy humans. Am J Clin Nutr. 2006 Sep;84(3):561-9. doi: 10.1093/ajcn/84.3.561. PMID 16960170